CLINICAL TRIAL: NCT02172963
Title: A Pilot Study Using Placenta Derived Decidual Stromal Cells for Hemorrhagic Cystitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olle Ringdén, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSCHC001
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hemorrhagic Cystitis
Keywords: Stem Cell Transplantation; Decidual Stromal Cells
MeSH Terms: conditions — Cystitis, Hemorrhagic

ARMS (1):
- Decidual Stromal Cell therapy for Hemorrhagic Cystitis (Experimental)
  Interventions: Biological: Decidual Stromal Cell therapy

INTERVENTIONS:
Biological: Decidual Stromal Cell therapy — Intravenous injection with placenta derived Decidual Stromal Cells. 1-2x10^6 cells/kg.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy using placenta derived decidual stromal cell therapy for hemorrhagic cystitis after allogeneic hematopoietic cell transplantation. It is hypothesized that the decidual stromal cell therapy is safe to infuse and that they have a positive clinical effect.

DETAILED DESCRIPTION:
Patients with grade 2-4 hemorrhagic cystitis will receive decidual stromal cell therapy at approximately 1-2x10^6 cells/kg once or at weekly intervals dependent on clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* Hemorrhagic cystitis grade 2-4

Exclusion Criteria:

* Urinary urge without macroscopic hematuria or clots

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response at day 28 after onset of hemorrhagic cystitis | 28 days after inclusion
  Disappearance of macroscopic hematuria.

SECONDARY OUTCOMES:
Actuarial survival at one year after onset of hemorrhagic cystitis | One year after inclusion
Time to disappearance of pain or urges | Up to 6 months after inclusion
Time to disappearance of microscopic hematuria | Up to 84 days after inclusion
Transplant related mortality | Up to one year after inclusion
  All mortality except for relapse
Incidence of severe infections | Up to one year after inclusion
  Incidence of severe bacterial, viral or fungal infections.
Incidence of graft versus host disease | Up to one year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringdén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden